CLINICAL TRIAL: NCT05208177
Title: A Phase Ⅰb/Ⅱ Dose-exploration and Efficacy-expansion Study of SHR-1802 Combined With Camrelizumab for Injection and Famitinib Malate Capsules for the Treatment of Advanced Solid Tumor
Brief Title: A Study of SHR-1802 in Patients With Advanced Solid Tumor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Adjustment of R&D strategy
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1802-II-201
Record Dates: First submitted 2022-01-18; First posted 2022-01-26 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — famitinib

STUDY DESIGN:
Intervention Model Description: Dose-escalation: Traditional 3+3 dose-escalation design. Dose-expansion: 10 to 12 subjects (included subjects of the dose-escalation part) will be enrolled in each tolerable dose level.
  Efficacy-expansion: After determination of the recommended dose for Phase II (RP2D), selected cohorts with different tumor types will be expanded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1802 for injection combined with Camrelizumab for Injection and Famitinib Malate Capsules (Experimental)
  Interventions: Drug: SHR-1802＋camrelizumab + famitinib

INTERVENTIONS:
Drug: SHR-1802＋camrelizumab + famitinib — SHR-1802 for injection，q3w； Camrelizumab for injection, q3w; Famitinib malate capsules, qd.

SUMMARY:
To assess the safety and tolerability of SHR-1802 combined with camrelizumab and famitinib in subjects with advanced solid tumor and to determine the dose-limiting toxicity (DLT)，recommended phase II dose (RP2D) and assess objective response rate (ORR) assessed by the investigator based on RECIST v1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
3. Has a life expectancy≥ 3 months;
4. At least one measurable lesion according to RECIST v1.1;
5. Pathologically confirmed advanced solid tumor;
6. Adequate bone marrow reserve and organ function.

Exclusion Criteria:

1. Have received prior therapy with camrelizumab, and famitinib;
2. Received anti-tumor therapies such as chemotherapy, radiotherapy, biological therapy, targeted therapy, or immunotherapy within 4 weeks before the first dose of the treatment;
3. Underwent a major surgery other than diagnosis or biopsy within 4 weeks before the first dose of the treatment;
4. Have uncontrolled clinically symptomatic pleural effusion, pericardial effusion, or ascites;
5. Have known history of arterial/venous thrombosis within 6 months prior to the first dose of the treatment, such as cerebrovascular accidents, deep vein thrombosis and pulmonary embolism;
6. Grade II-IV cardiac insufficiency as per the New York Heart Association (NYHA) criteria; arrhythmia requiring long-term drug control; unstable angina or acute myocardial infarction within 6 months before the first dose of the treatment;
7. Have other potential factors that may affect the study results or result in the premature discontinuation as determined by the investigator, such as alcoholism, drug abuse, substance abuse, other serious diseases (including mental illness) requiring concomitant treatment, serious laboratory abnormalities, or family or social factors that could affect the safety of medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 4 weeks
Recommended phase II dose (RP2D) | up to 1 years
ORR | up to 2 years
  Objective Response Rate, determined according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
DOR | up to 2 years
  Duration of Response, determined according to RECIST v1.1 criteria
DCR | up to 2 years
  Disease Control Rate, determined according to RECIST v1.1 criteria
PFS assessed by investigator | up to 2 years
  Progression Free Survival, determined according to RECIST v1.1 criteria
TTR | up to 2 years
  Time to Response，determined according to RECIST v1.1 criteria
OS (overall survival) | up to 2 years
  From date of treatment start to any cause death or last follow-up
12-month OS rate | from the date of the first dose up to 2 years
AEs+SAEs | from the first drug administration to within 90 days for the last drug dose
  Adverse Events and Serious Adverse Events assessed by CTCAE v5.0
Concentration of drug in serum | 0.5 hour before the first dose up to 30 days after last dose
  Serum concentration of Camrelizumab for Injection and SHR-1802 for injection.
Concentration of drug in plasma | n the second cycle，predose 1 hour and 6 hours post-dose；In cycle 3, cycle 4, cycle 6, cycle 8, and cycle 10，predose 1 hour（each cycle is 21 days）
  Plasma concentration of Famitinib malate capsule and its metabolite.
Count of T lymphocyte subsets | 30 minutes before the first dose of SHR-1802, the 4th and 8th days after the first injection
  Count of CD4+ T lymphocyte subsets in peripheral blood；Count of CD8+ T lymphocyte subsets in peripheral blood.
Percentage of T lymphocyte subsets | 30 minutes before the first dose of SHR-1802, the 4th and 8th days after the first injection
  Percentage of CD4+ T lymphocyte subsets in peripheral blood；Percentage of CD8+ T lymphocyte subsets in peripheral blood.
ADA | up to 30 days after last dose
  Anti-drug antibody of Camrelizumab for Injection and SHR-1802 for injection
Nab | up to 30 days after last dose
  Neutralizing Antibody of Camrelizumab for Injection and SHR-1802 for injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute&Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided